CLINICAL TRIAL: NCT06800989
Title: To Assess the Contribution of Sophrology Assisted by an Ambulatory Device on the Anxiety of Patients Undergoing Chemotherapy for the Treatment of Localized Breast Cancer.
Acronym: DOMI-SOPHRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-2024-11
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Female
Keywords: anxiety; sophrology; breast cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a regional multicenter, controlled, randomized 2:1, prospective study. Stratification will be based on the center and age (< 50 years / ≥ 50 years)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sophrology + Morphée® device (Experimental): The Morphée® device is an easy-to-use ambulatory sophrology tool in French. Patients will be encouraged to perform at least one daily ambulatory sophrology session with the Morphée® device, according to a support plan defined with the sophrologist.
  Two sophrology sessions will be conducted in the experimental group. The first session (S1) should take place on Cycle 1 Day 1 or within a maximum of 3 weeks following Cycle 1 Day 1. The second session (S2) should be conducted within 3 to 4 weeks after the first session
- Standard of care (No Intervention): In the control arm, patients will be managed according to current recommendations, including information and access to support care available in the investigator centers.
  After participation in the study, patients may be offered a session of sophrology at the investigator's discretion.

INTERVENTIONS:
Behavioral: sophrology sessions — Two sophrology sessions will be conducted in the experimental group. The first session (S1) should take place on Cycle 1 Day 1 or within a maximum of 3 weeks following Cycle 1 Day 1. The second session (S2) should be conducted within 3 to 4 weeks after the first session.
Device: Morphee Device — Patients will be encouraged to perform at least one daily ambulatory sophrology session with the Morphée® device, according to a support plan defined with the sophrologist.

SUMMARY:
Patients with localized breast cancer undergo treatment that includes breast surgery, which always alters their body image, complemented by optional additional treatments depending on the specifics and severity of their disease. These treatments are multimodal and may include chemotherapy, radiotherapy, targeted anticancer treatments, and hormone therapy, followed by prolonged monitoring for at least 5 years.

A recent study showed that the announcement of cancer and its treatments is a source of reactive anxiety for 47% of patients at the time of diagnosis, which can be associated with depression in 59% of cases before chemotherapy. Anxiety increases with the intensity of treatments and is higher when chemotherapy is administered, especially in younger patients (under 50 years old).

The integrative multidisciplinary care available in treatment centers (psychologist, adapted physical activity, socio-aesthetician), combined with external support through associative networks (art therapy, music therapy, etc.), is crucial for improving quality of life and treatment side effects. Sophrology is one of these complementary therapies recommended by Association Francophone Des Soins Oncologiques De Support (French Association for Supportive Care in Oncology) within or outside the healthcare structure and is validated as supportive care. Its principle is to positively enhance patients' qualities and resources by altering states of consciousness, allowing individuals to find a balance between their thoughts, emotions, and behaviors. The three fundamental principles are to bring the body schema to a more lived reality, reinforce positive action, and develop objective reality. The "mindfulness" techniques used in sophrology include dynamic relaxation and sophronizations. Sophrology is based on the scientific principles of mindfulness meditation (developing attentional resources and body awareness by modulating brain waves).

Studies have shown the benefits of mindfulness in managing stress, certain psychosomatic conditions, and chronic pain. Improvements in overall quality of life, stress symptoms, and sleep quality have been reported in the evaluation of a mindfulness meditation program for cancer patients. A trial demonstrated the beneficial effect of group mindfulness meditation on the anxiety of women who had undergone chemotherapy for breast cancer.

Today, although sophrology is regularly used in medical care, no robust scientific study has evaluated its benefit in oncology. Institut National de la Santé et de la Recherche Médicale, together with Haute Autorité de la Santé, highlighted in its 2020 report on sophrology the significant need to scientifically assess the interest of sophrology in medical care.

However, the use and accessibility of complementary therapies, including sophrology, are very unequal across France and depend on hospitals, geography, patient mobility, and sometimes the financial ability of patients to access paid complementary therapies. As a result, many anxious patients cannot access sophrology sessions at the desired time due to geographical, accessibility, human resource, and sometimes financial reasons (outside the hospital).

The Morphée® device could help reduce these disparities and accessibility issues by allowing patients to perform a sophrology session at any time and place after receiving explanations from a healthcare professional.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with localized breast cancer
2. Patient > 18 years old
3. Patient requiring chemotherapy +/- combined with immunotherapy or targeted therapy, in neoadjuvant or adjuvant seeting defined by the multidisciplinary consultation meeting.
4. Patient with signed consent
5. Patient has national health insurance coverage

Exclusion Criteria:

1. Patient previously treated with chemotherapy for breast cancer
2. Patient with metastatic breast cancer
3. History of psychiatric illness or treatment with neuroleptics, antidepressants or thymoregulators thymoregulator, prior to discovery of cancer (except resolved depressive episode, without psychiatric treatment for at least 2 years). An anxiolytic or hypnotic treatment prescribed after diagnosis is authorized
4. Patient suffering from psychiatric disorders, delusional phases, schizophrenia contraindicating practice of sophrology
5. Patient who has already had an introduction to sophrology in the context of her pathology, or who plans to start sophrology within within 3 months of the start of treatment outside the hospital structure and by her own means
6. Patient does not understand or speak French
7. Cognitive impairment or inability to understand, compromising participation in the study and use and understanding of the device
8. Patient under legal protection, guardianship or trusteeship
9. Inability to undergo protocol monitoring for geographical or social reasons.
10. Patient participating in another interventional study evaluating supportive care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
To measure the evolution of anxiety in patients undergoing adjuvant or neoadjuvant chemotherapy treatment, depending on whether they benefit from a sophrology program through an ambulatory sophrology device (Morphée®) | Inclusion and 3 months after start of treatment
  Anxiety evaluated with Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains

CONTACTS AND LOCATIONS:
Overall Officials: Simmet, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (3):
- France (3):
  - Institut de Cancérologie de l'Ouest - site Angers, Angers
  - CH Cholet, Cholet
  - Institut de Cancérologie de l'Ouest - site Saint Herblain, Saint-Herblain